CLINICAL TRIAL: NCT04742166
Title: Impact of Side to Side Gastrojejunostomy on the Rate of Delayed Gastric Emptying After Pancreaticoduodenectomy: A Prospective Randomized Study
Brief Title: Impact of Side to Side Gastrojejunostomy on the Rate of Delayed Gastric Emptying After Pancreaticoduodenectomy (IPAD)
Acronym: IPAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC20_8891_IPAD Study
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Surgical Technique
MeSH Terms: interventions — Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Side to side gastrojejunal reconstruction (Experimental): The post-operative care: usual practise Follow-up: 90 days postoperatively
  At Day 90:
  * a blood test for albumin and prealbumin
  * a GIQLI questionnaire (quality of life score) to be completed by the patient
  Interventions: Procedure: Reconstruction
- Terminolateral gastrojejunal reconstruction (Active Comparator): The post-operative care: usual practise Follow-up: 90 days postoperatively
  At Day 90:
  * a blood test for albumin and prealbumin
  * a GIQLI questionnaire (quality of life score) to be completed by the patient
  Interventions: Procedure: Reconstruction

INTERVENTIONS:
Procedure: Reconstruction — Lateral gastrojejunal Terminolateral gastrojejunal

SUMMARY:
Prospective bi-centric randomized open-label study comparing side to side and end to side gastrojejunostomy in pancreaticoduodenectomy

DETAILED DESCRIPTION:
Delayed gastric emptying is one of the main complications occurring after pancreatodudodenectomy, the incidence of which is estimated between 10 and 40% in the literature. Its occurrence leads to an alteration in post-operative quality of life (maintenance or resting of the nasogastric tube) and is the primary reason an increase in the length of hospital stay and therefore the cost of treatment. In addition, it predisposes to the risk of inhalation pneumopathy, which increases the risk of post-operative death. Various technical surgical points have been suggested by retrospective studies to reduce its incidence (pyloric preservation, respect for the left gastric vein, ante-colic positioning of the Child's handle, making a Y-shaped handle) but without ever being validated in randomized prospective studies.

Recently three retrospective studies have highlighted the interest of performing a side to side l rather than an end to side gastro-jejunal anastomosis to reduce the rate of post-operative delayed gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years old
* to benefit from a cephalic duodenopancreatectomy whatever the indication (benign and malignant tumor)
* affiliated with a health insurance system
* having received oral and written information about the protocol and having signed a free and informed written consent.

Exclusion Criteria:

* associated organ resection except for portal vein or hepatic artery resection.
* history of gastric or esophageal resection
* person subject to legal protection (safeguard justice, trusteeship and guardianship) and persons deprived of liberty
* pregnant or breastfeeding women
* patient participating in another clinical trial that may interfere with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative delayed gastric emptying | Day 90
  Occurrence of post-operative delayed gastric emptying (classified to the International Study Group for Pancreatic Surgery (ISGPS))

SECONDARY OUTCOMES:
Occurrence of Clavien-Dindo complications | Up to day 90
Pancreatic fistula | Up to day 90
  Occurence of pancreatic fistula (classified according to the ISGPS classification)
Biliary fistula | Up to day 90
  Occurrence of biliary fistula
Haemorrhage | Up to day 90
  Occurrence of haemorrhage according to the ISGPS classification
Food intake (liquid and solid) | Up to five days after surgery
  Time to oral food intake
First gas | Up to five days after surgery
  Time to the emission of the first gas
Pre-operative to 3-month post-operative weight ratio | Up to day 90
Albumin and prealbumin levels | Up to day 90
General Quality of Life Score for Digestive Pathologies | Up to day 90
Gastrointestinal Quality of Life Index (GIQLI) | Up to day 90
Mortality rate | Day 30
Mortality rate | Day 90
Time to functional recovery (days) after surgery | Day 90
  Functional recovery defined as all of the following:
  * independently mobile at the preoperative level
  * sufficient pain control with oral medication alone
  * ability to maintain at least 50% daily required caloric intake
  * no intravenous fluid administration
  * no clinical signs of infection when other criteria were met

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Paoli Calmettes, Marseille
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No